CLINICAL TRIAL: NCT03208114
Title: Does the Information on Breast Milk Substitutes at Hospital Discharge Affect Breastfeeding Behavior at Six Months? A Randomized Controlled Trial
Brief Title: Information on Breast Milk Substitutes at Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Discharge_RCT
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-07

CONDITIONS: Breastfeeding
Keywords: breastfeeding, support, promotion
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A total mother-infant pairs enrolled will be randomized to either receive the written information of the name of a breast milk substitute on the infant's discharge documents (group A) or not to receive it (group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Receiving the written information of the name of a breast milk substitute on the infant's discharge documents
  Interventions: Other: Receiving written information on breast milk substitute
- Group B (No Intervention): Not receiving the written information of the name of a breast milk substitute on the infant's discharge documents

INTERVENTIONS:
Other: Receiving written information on breast milk substitute — Receiving written information on breast milk substitute
  Arms: Group A

SUMMARY:
Background: Although exclusively breastfeeding is recommended up to six months, current breastfeeding rates are still far from recommended targets. The investigators aim to investigate the effect of the information on breast milk substitutes at discharge on breastfeeding rates at six months of age.

Methods: A randomized controlled trial has been designed. All mother-infant pairs will be randomized to either receive the written information of the name of a breast milk substitute on the infant's discharge documents (group A) or not to receive it (group B). Mothers will receive a phone interview on mode of infants' feeding at 7 days,1, 2 , 3 and 6 months after delivery. Reasons for early discontinuation of breastfeeding according to mothers' opinion will be also collected.

Statistical analysis:

Sample size: In order to detect a 10% difference in the discontinuation rate of exclusive breastfeeding at six months of age between groups, at 5% significance and 80% power, a total of 388 mother-infant pairs per group will need.

Descriptive data will be expressed as mean±SD or number of observations (percentage). With regard to the items that were scored on a 5-point Likert scale, for the analysis, the answers will categorize into two groups (not important and important).

Differences between groups in breastfeeding rates at each time point of the study will be assessed by the T-test analysis. The X2 test will be used for comparisons between discrete variables. Statistical significance is set at a = .05 level. All statistical analyses will be performed by using SPSS (version 12, SPSS, Chicago, IL).

DETAILED DESCRIPTION:
Background: To investigators' knowledge there is paucity of data regarding the effect of the information of breast milk substitutes written on newborn's discharge medical documents on subsequent breastfeeding behavior.

The aim of the study is to investigate the effect of the information of breast milk substitutes written on newborn's discharge documents on breastfeeding rates at six months of age in a cohort of mothers exclusively breastfeeding at hospital discharge. The hypothesis to be tested is that the breastfeeding rates of the mothers receiving the written information of the name of a breast milk substitute at discharge would be similar to that of the breastfeeding mothers not receiving it.

Methods

Ethics Statement

The study was approved by the Ethics Committee of the Fondazione Istituto di Ricovero e Cura a Carattere Scientifico Cà Granda Ospedale Maggiore Policlinico, and informed written consent will be obtained from the parents.

Design

The investigator will conduct a prospective, controlled, single-blinded randomized trial. Breastfeeding will be promoted and supported in all mother-infant pairs throughout hospital stay. Enrollment and randomization will occur concurrently at discharge. Mother-infant pairs will be randomized either to receive the written information of the name of a breast milk substitute on the infant's discharge documents (group A) or not to receive it (group B). Randomization to group A or B will be performed by an independent investigator with a random permuted block size of 4.

Procedures

At enrollment the following maternal variables will be collected through a face to face interview: mode of delivery (vaginal delivery/caesarean section), being primiparous or multiparous, previous breastfeeding experience (yes/no; if yes how many days/months), labour duration, drugs consumption during pregnancy and/or labour, including analgesia or anesthesia, diseases arisen during pregnancy, maternal education classified as low (≤13 years) or high (>13 years), pre and post pregnancy body mass index (kg/m2), marital status, age and attitude towards smoking. Mothers will be also interviewed on pre pregnancy course attendance, intention to breastfeed and satisfaction with the breastfeeding support received during hospital stay. Timing of the first latching will be also registered.

The following neonatal variables will be also collected: gestational age, gender, Apgar score values at 1 and 5 minutes, birth weight, length and head circumference.

Mothers will be contacted at 7 (±3) days,1 (±7 days), 2 (±7 days), 3 (±7 days), 6 (±7 days) months after delivery by phone calls by four investigators blinded to randomization. Following a structured interview mothers will be asked whether the infant had been breastfed during the last 24 hours. Mothers will be then asked whether the infant had been fed any water and/or fruit juice and/or formula and/or semi solid and/or solid foods during the last 24 hours.

Mode of feeding (exclusive breastfeeding, predominant breastfeeding, mixed breastfeeding exclusive formula feeding) will be then categorized according to the World Health Organization.

If the infant will be no more breastfed, mothers will be administered a questionnaire modified after Odom et al. in order to investigate the main reasons associated with breastfeeding discontinuation. Specifically, the questionnaire focuses on the following 7 macro areas: lactation problems, milk-pumping factors, psychosocial factors, nutritional factors, life style factors, medical problems, factors related to the infant.

Mothers will be asked to rate the importance of each item of the questionnaire according to a 5-point Likert scale: score 1=not at all important, score=2=not very important, score=3 moderately important, score=4 important, score=5 extremely important.

Adverse events

Adverse events will be assessed based on inquiries to the mothers. All adverse events will be evaluated by the investigator for severity. An adverse event will be defined as any event that will not be consistent with the information provided in the consent form or that could not reasonably be expected to accompany the natural history and progression of the subject's condition throughout the study. Adverse events will be considered serious if fatal or life-threatening, require hospitalization or surgical intervention, result in persistent or significant disability/incapacity or are considered to be medically relevant by the investigator. All other adverse events will be categorized as non-serious.

Statistical analysis

Sample size

In order to detect a 10% difference in the discontinuation rate of exclusive breastfeeding at six months of age between groups, at 5% significance and 80% power, a total of 388 mother-infant pairs per group were needed.

Descriptive data will be expressed as mean±SD or number of observations (percentage). With regard to the items that are scored on a 5-point Likert scale, for the analysis, the answers will be categorized into two groups (not important and important).

Differences between groups in breastfeeding rates at each time point of the study will be assessed by the T-test analysis. The X2 test will be used for comparisons between discrete variables. Statistical significance will be set at a = .05 level. All statistical analyses will be performed by using SPSS (version 12, SPSS, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Birth weight > 2500 g
* Gestational age ≥ 37 weeks
* Singleton pregnancy
* Being exclusively breastfed from birth to discharge
* Caucasian race

Exclusion Criteria:

* presence of congenital diseases
* presence of chromosomal abnormalities
* presence of perinatal infections
* presence of cardio-respiratory instability
* being born to mothers affected by endocrine and/or metabolic and/or gastrointestinal and/or renal diseases.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 802 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding rates. | Six months of life
  Evaluation of exclusive breastfeeding rates according to randomization's group.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Mosca, Prof, Principal Investigator — NICU. Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano, Milan, Italy, 20122

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartick MC, Jegier BJ, Green BD, Schwarz EB, Reinhold AG, Stuebe AM. Disparities in Breastfeeding: Impact on Maternal and Child Health Outcomes and Costs. J Pediatr. 2017 Feb;181:49-55.e6. doi: 10.1016/j.jpeds.2016.10.028. Epub 2016 Nov 10. PMID 27837954
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Rollins NC, Bhandari N, Hajeebhoy N, Horton S, Lutter CK, Martines JC, Piwoz EG, Richter LM, Victora CG; Lancet Breastfeeding Series Group. Why invest, and what it will take to improve breastfeeding practices? Lancet. 2016 Jan 30;387(10017):491-504. doi: 10.1016/S0140-6736(15)01044-2. PMID 26869576
- [Background] Mason F, Rawe K, Wright S. Superfood for Babies: How Overcoming Barriers to Breastfeeding will Save Lives. London: Save the Children; 2013.
- [Background] Baker P, Smith J, Salmon L, Friel S, Kent G, Iellamo A, Dadhich JP, Renfrew MJ. Global trends and patterns of commercial milk-based formula sales: is an unprecedented infant and young child feeding transition underway? Public Health Nutr. 2016 Oct;19(14):2540-50. doi: 10.1017/S1368980016001117. Epub 2016 May 23. PMID 27211798
- [Background] McFadden A, Mason F, Baker J, Begin F, Dykes F, Grummer-Strawn L, Kenney-Muir N, Whitford H, Zehner E, Renfrew MJ. Spotlight on infant formula: coordinated global action needed. Lancet. 2016 Jan 30;387(10017):413-5. doi: 10.1016/S0140-6736(16)00103-3. No abstract available. PMID 26869552
- [Background] Piwoz EG, Huffman SL. The Impact of Marketing of Breast-Milk Substitutes on WHO-Recommended Breastfeeding Practices. Food Nutr Bull. 2015 Dec;36(4):373-86. doi: 10.1177/0379572115602174. Epub 2015 Aug 27. PMID 26314734
- [Background] Sobel HL, Iellamo A, Raya RR, Padilla AA, Olive JM, Nyunt-U S. Is unimpeded marketing for breast milk substitutes responsible for the decline in breastfeeding in the Philippines? An exploratory survey and focus group analysis. Soc Sci Med. 2011 Nov;73(10):1445-8. doi: 10.1016/j.socscimed.2011.08.029. Epub 2011 Sep 17. PMID 21978633
- [Background] Odom EC, Li R, Scanlon KS, Perrine CG, Grummer-Strawn L. Reasons for earlier than desired cessation of breastfeeding. Pediatrics. 2013 Mar;131(3):e726-32. doi: 10.1542/peds.2012-1295. Epub 2013 Feb 18. PMID 23420922
- [Derived] Mosca F, Roggero P, Garbarino F, Morniroli D, Bracco B, Morlacchi L, Mallardi D, Gianni ML, Consonni D. Determinants of breastfeeding discontinuation in an Italian cohort of mother-infant dyads in the first six months of life: a randomized controlled trial. Ital J Pediatr. 2018 Nov 6;44(1):134. doi: 10.1186/s13052-018-0572-z. PMID 30400806
- See also: The link refers to a book on the global strategy for infant and young child feeding — http://whqlibdoc.who.int/publications/2003/9241562218.pdf